CLINICAL TRIAL: NCT03739827
Title: Natural History and Biospecimen Acquisition Study for Children and Adults With Rare Solid Tumors
Brief Title: Natural History and Biospecimen Acquisition for Children and Adults With Rare Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190016; 19-C-0016
Record Dates: First submitted 2018-11-10; First posted 2018-11-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-07-24

CONDITIONS: Malignant Solid Tumors; Other Neoplasms Solid Tumors; Pediatric Solid Tumor; Refractory Solid Tumors; Solid Tumor
Keywords: Service to the Patients; Knowledge about the Nature of Cancer; Cancer Evaluations; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1/Cohort 1: Subjects with a diagnosis of rare tumor (fewer than 15 cases in 100,000 people per year)
- 2/Cohort 2: Relatives of subjects with a rare tumor who have a germline genetic variant that predispose to a rare solid tumor or a subject who has a germline genetic variant that predispose to a rare solid tumor
- 3/Cohort 3: Relatives of subjects with a diagnosis of rare tumor that do NOT have known germline genetic variants that predispose to a rare solid tumor.
- 4/ Cohort 4: Parents/guardians of children with a diagnosis of rare tumor participating in focus groups (if not enrolled in Cohorts 1, 2 or 3)

SUMMARY:
Background:

Approximately 150 cases of cancer per one million per year are considered rare cancers. While all tumors originate from genetic changes, a small percentage of these tumors are familial. Researchers want to study these changes in biological samples from people with rare tumors in order to learn more about how these tumors develop. The information obtained from this study may lead to improved screening, preventive guidelines, and treatments.

Objective:

To better understand rare cancers and hereditary cancer syndromes.

Eligibility:

People who have a rare tumor, a family history of a rare tumor, a hereditary cancer syndrome, or a mutation that leads to rare tumors.

Design:

Participants will be screened with questions about their medical history and/or that of their family members. They will give a saliva sample.

Participants who have a tumor will have their medical records and tests reviewed. They will answer questions about their wellbeing and needs. They may provide a tumor tissue sample.

Participants may also have:

* Physical exam
* Clinical photography
* Blood, urine, saliva, and stool samples taken
* Consultation with specialists
* A scan that produces a picture of the body. Either one that uses a small amount of radiation, or one that uses a magnetic field.
* Genetic testing/genetic counseling.

Participants will be contacted once a year. They will answer updated questions about their medical and family history.

Participants will be asked to contact the study team if there are changes in their tumors.

Participants may be invited to join focus groups for people with the same diagnosis of rare tumors.

Participants may be invited to participate in other NIH protocols.

****************************************

****************************************

RARE TUMOR LIST:

1. Acinar cell carcinoma of the pancreas
2. Adamantinoma
3. Adenosqaumous carcinoma of the pancreas
4. Adrenocortical carcinoma
5. Alveolar soft part sarcoma
6. Anaplastic Thyroid Cancer
7. Angiosarcoma
8. Atypical Teratoid Rhabdoid Tumor/MRT
9. Carcinoid
10. Carcinoma of Unknown Primary
11. Chondrosarcoma
12. Chondromyxoid fibroma
13. Chordoma
14. Clear cell renal carcinoma
15. Clear Cell Sarcoma
16. Clear cell sarcoma of kidney
17. Conventional chordoma
18. Dedifferentiated chordoma
19. Desmoid
20. Desmoplastic small round cell tumor
21. Epithelioid hemangioendothelioma
22. Esthenioneuroblastoma
23. Ewing Sarcoma
24. Fibrolamellar carcinoma
25. Fusion negative rhabdomyosarcoma
26. Fusion positive renal cell carcinoma
27. Fusion positive rhabdomyosarcoma
28. Gastro-enteropancreatic neuroendocrine tumor
29. Hepatoblastoma
30. Hereditary Diffuse Gastric Cancer
31. Inflammatory myofibroblastic tumor
32. Kaposiform hemangioendothelioma
33. Malignant ectomesenchymal tumor
34. Malignant peripheral nerve sheath tumor
35. Malignant triton tumor
36. Medullary thyroid cancer
37. Mixed acinar adenocarcinoma
38. Mixed acinar neuroendocrine carcinoma
39. Myxoid Liposarcoma
40. Neuroblastoma
41. Neuroendocrine tumors
42. NUT midline carcinoma
43. Osteosarcoma
44. Pancreas ductal adenocarcinoma with squamous features
45. Pancreatic acinar cell carcinoma
46. Papillary renal cell carcinoma
47. Paraganglioma
48. Parosteal Osteosarcoma
49. Periosteal Osteosarcoma
50. Peripheral nerve sheath tumor
51. Peripheral primitive neuroectodermal tumor
52. Pheochromocytoma
53. Pituitary cancer
54. Poorly differentiated chordoma
55. Renal medullary carcinoma
56. Rhabdomyosarcoma
57. Round cell Liposarcoma
58. Schwannoma
59. Sclerosing Epithelioid Fibrosarcoma
60. SDH deficient GIST
61. SMARCB1 deficient tumors
62. SMARCA4 deficient tumors
63. Synovial sarcoma
64. Undifferentiated Sarcoma

    ****************************************

    ****************************************

DETAILED DESCRIPTION:
Background:

Rare tumors are defined as fewer than 150 incident cases per one million per year. Consequently, only 11 tumor types are common in U.S. adults (prostate, breast, lung/bronchus, colon, uterus, bladder, melanoma, rectum, ovary, non-Hodgkin lymphoma, and kidney/renal pelvis neoplasms) and will not be studied in this trial. One-quarter of all adults with tumor have a rare tumor diagnosis.

All pediatric tumors meet this definition of rare affecting < 1% individuals younger than 20 years per year in the US.

Notably, there is a group of solid tumors that occur so infrequently in children and adults that little is known about the natural history of these tumors, their clinical behavior, molecular/genetic characteristics, optimal management, and drug response.

The NCI and the NIH Clinical Center infrastructure are uniquely suited to conduct studies of rare tumors. There is a precedent in the NCI when even non-interventional studies or initiatives were paradigm-changing. The NCI neurofibromatosis type 1 natural history study allowed the development of groundbreaking interventional trials in participants with plexiform neurofibromas. The Pediatric and Wild-Type Gastrointestinal Stromal Tumor (GIST) Clinic, which involves intramural and extramural experts, not only provided the background for discovery of the molecular features of a very rare disease such as succinate dehydrogenase deficient GIST, but also was able identify therapeutic strategies for this group of participants (for example, avoidance of unnecessarily aggressive surgery). Similarly, studies in adults at the CCR have tremendously advanced the understanding of rare solid tumors occurring primarily in adults such as thymoma, renal cell cancer, and endocrine tumors.

Systematic and longitudinal collection and annotation of clinical history, tissue samples, imaging studies, patient reported outcomes, and other pertinent information in participants with these rare tumors and return of results to participants will provide a service to the participants themselves and to the medical community, in line with the NIH mission of to seek fundamental knowledge about the nature and behavior of living systems and the application of that knowledge to enhance health, lengthen life, and reduce illness and disability .

Objective:

To comprehensively and longitudinally evaluate the natural history of participants with rare solid tumors or tumor predisposition syndromes, estimating and defining their clinical spectrum (e.g. disease course and survival).

Eligibility:

Participants with a diagnosis of a rare solid tumor (fewer than 15 cases in 100,000 people per year).

OR

Relatives of participants with diagnosis of rare solid tumors

OR

Carriers of germline genetic variants that predispose to rare solid tumor and their relatives.

Design:

This will be a long-term study to comprehensively study participants (and their relatives) with select rare tumors.

Initially participants will provide clinical information (medical history, family medical history, imaging studies and reports, surgical pathology reports, genetic test results, patient-reported outcomes) and biospecimens (archival pathology specimen and saliva) for review by and feedback from the study team.

If indicated, participants will be invited to the study site for additional evaluations and consultation, including clinical phenotyping, genotyping, imaging of tumor sites, and patient reported or other appropriate outcomes.

After evaluation, participants will be provided with recommendations about possible treatment options and might be enrolled into disease specific sub-protocols of this trial.

Since long-term follow-up of individuals with rare tumors, their family members at high risk for developing tumors, and carriers of germline genetic variants is a major feature of the study, we intend to maintain active contact with study subjects for as long as possible.

In addition to evaluating individual participants, this protocol will allow bringing groups of participants (approximately 10-20) with specific rare tumors for a rare tumor clinic on the same day to allow for development of a deeper understanding of rare tumors through the conduct of focus groups.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Cohort 1: Participants with a diagnosis of a rare solid tumor (fewer than 15 cases in 100,000 people per year). There are no age restrictions beyond the neonatal period (4 weeks).

OR

-Cohort 2: Participants without a rare tumor who have a germline genetic variant that predisposes to a rare solid tumor

OR

-Cohort 3: Relatives of participants with diagnosis of rare solid tumors who do NOT have a known germline variant that predisposes to a rare solid tumor

OR

* Cohort 4: Parent/guardian of child participating in a focus group if not already enrolled on the study.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

None

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
To comprehensively and longitudinally evaluate the natural history of patients with rare solid tumors or tumor predisposition syndromes, estimating and defining their clinical spectrum (e.g. disease course and survival) | 10 years
  To comprehensively and longitudinally evaluate the natural history of patients with rare solid tumors or tumor predisposition syndromes, estimating and defining their clinical spectrum (e.g. disease course and survival)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Wedekind Malone, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Oregon Health and Science University, Portland, Oregon
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0016.html